CLINICAL TRIAL: NCT05811611
Title: Efficacies of Two WeChat Mini Program-based Interventions in Reducing Sexual Risk Behaviors Among Heterosexual Male Factory Workers in China: a Randomized Controlled Trial
Brief Title: Two WeChat Mini Program-based Interventions Reducing Sexual Risk Behaviors Among Heterosexual Male Factory Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HLPM201907020105
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Behavior, Sex
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WeChat Mini Program plus tailored online promotion videos (Experimental): 1. Having access to a WeChat Mini Program providing HIV and STI prevention information during the project period
  2. The WeChat Mini Program proactively asks questions assessing sexual risk behaviors at Month 0 and Month 1, and invite participants two watch online health promotion videos tailored to their sexual risk behaviors status.
  Interventions: Behavioral: WeChat Mini Program plus tailored online health promotion videos
- WeChat Mini Program Only (Active Comparator): Having access to a WeChat Mini Program providing HIV and STI prevention information during the project period
  Interventions: Behavioral: WeChat Mini Program Only

INTERVENTIONS:
Behavioral: WeChat Mini Program plus tailored online health promotion videos — Participants have access to a WeChat Mini Program. Participants will also watch online health promotion videos tailored to their current sexual behaviors.
  Arms: WeChat Mini Program plus tailored online promotion videos
Behavioral: WeChat Mini Program Only — Participants only have access to a WeChat Mini Program.
  Arms: WeChat Mini Program Only

SUMMARY:
A non-blinded parallel group randomized controlled trial is conducted. Adult male full-time employees of factories in Shenzhen who have access to smartphone and WeChat are recruited by staff of the Longhua Center for Disease Control and Prevention (CDC).

After completing an online baseline questionnaire, participants will be randomized evenly to either the intervention group or the control group. Participants in the control group will have access to a WeChat Mini Program providing HIV and sexually transmitted prevention information during the project period. In addition to those received by the control group, the Mini Program will proactively ask participants in the intervention group some simple questions to assess presence of sexual risk behaviors at Month 0 and Month 1, and invite them to watch online health promotion video(s) tailored to their current sexual risk behaviors.

All participants will complete two online follow-up surveys six and twelve months after completion of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male at birth
* Aged 18 years or above
* Full-time employee of a factory in Shenzhen
* Having a smartphone with internet access
* Having installed or willing to install WeChat on the smartphone
* Willing to complete follow-up surveys at Month 6 and 12

Exclusion Criteria:

* Oral or anal sex with a man
* Blindness ot deafness
* Not able to communicate effectively with project staff
* Self-reported as HIV positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male at birth
Enrollment: 244 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Sexual intercourse with non-regular female sex partner | 6 months
  Proportion of the participants who have sexual intercourse with a non-regular female sex partner in the past six months
Sexual intercourse with female sex workers | 6 months
  Proportion of participants who have sexual intercourse with a female sex worker in the past six months

SECONDARY OUTCOMES:
Condomless sex with non-regular female sex partners | 6 months
  Proportion of the participants who have condomless sex with a non-regular female sex partner in the past six months
Condomless sex with female sex workers | 6 months
  Proportion of the participants who have condomless sex with a female sex worker in the past six months

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data involve sensitive sexual behaviors of the participants

REFERENCES:
- [Derived] Zhang K, Cao B, Fang Y, Liang X, Ye D, Chen YQ, Zhong R, Cao H, Hu T, Li T, Cai Y, Zou H, Wang Z. Comparing the Efficacy of 2 WeChat Mini Programs in Reducing Nonmarital Heterosexual Contact by Male Factory Workers: Randomized Controlled Trial. J Med Internet Res. 2024 Sep 9;26:e49362. doi: 10.2196/49362. PMID 39250213